CLINICAL TRIAL: NCT01454362
Title: Phase 4 Study to Compare of the Effects of the Electronic Cigarette and Nicotine Inhalator on Tobacco Withdrawal Symptoms Over 24 Hours of Abstinence
Brief Title: Effect of the Electronic Cigarette on Withdrawal Symptoms
Acronym: ECIG24
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Hayden McRobbie, Reader in Public Health Interventions, Queen Mary University of London
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: QMUL111111; 2011-005565-20 (EudraCT Number); U1111-1127-4445 (Other: WHO: Universal Trial Number (UTN))
Record Dates: First submitted 2011-10-12; First posted 2011-10-19 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Mental and Behavioral Disorders; Withdrawal State
Keywords: nicotine; inhalator; electronic cigarette; tobacco
MeSH Terms: conditions — Mental Disorders; Vaping | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electronic cigarette (Experimental): We analysed 15 brands of the most popular E-Cs in the UK, EU and US for nicotine levels in the mist. Vapours were generated from cartridges of various nicotine content using a standard single-port linear smoking machine with a puff volume of 70 ml, 1 puff every 7 sec., and a puff duration of 1.8 sec (based on averaged puffing conditions from 10 E-C users found during preliminary studies). Nicotine was absorbed in two sequential washing bottles with methanol and internal standards and analysed with gas chromatography. One brand was selected for this study as it consistently delivers about 1mg of nicotine with 20 puffs.
  Interventions: Drug: Nicotine
- Nicotine Inhalator (Active Comparator): The inhalator consists of a nicotine cartridge which is placed into a plastic mouthpiece. One cartridge contains 10mg of nicotine of which 4mg of nicotine can be extracted. Nicotine is delivered mainly through the oral cavity, throat, and upper respiratory tract with a minor fraction reaching the lungs. A single cartridge can be used for one 20-minute period of continuous puffing or periodic use of up to 400 puffs per cartridge.
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Inhalation of nicotine.
  Other Names: Nicorette inhalator

SUMMARY:
Study rationale: Sensory/behavioural elements of smoking play a role in smoking behaviour and may have a potential to assist smoking cessation. Among current treatments for smokers, only the nicotine inhalator is attempting to address such factors. The inhalator's efficacy does not exceed that of the other nicotine replacement therapy (NRT) products, but it mimics the relevant sensory input to only a limited extent, and its nicotine delivery is dependent on intensive puffing. Recently a new product, the Electronic Cigarette (E-C) has become available, which provides a more realistic behaviour and sensory replacement for smoking and can provide good nicotine levels with less effort.

Primary objective: To compare E-C and nicotine inhalator in their effects on tobacco withdrawal symptoms over 24hr abstinence.

Hypotheses: E-C will be more effective than the inhalator in reducing withdrawal symptoms and craving and elicit more favorable user ratings. It will also provide higher nicotine levels.

Study design: In a cross-over study, participants will be randomized to the sequence of conditions and provide baseline measures and samples for salivary cotinine analysis. They will be asked to abstain from smoking their usual cigarettes and use the allocated product over 24 hours. They will return to the study centre the following day, and complete measures of craving and withdrawal, ratings of subjective and sensory effects of the products, product satisfaction, and adverse effects. They will also provide saliva samples for cotinine analysis. Abstinence from smoking will be verified with CO readings.

DETAILED DESCRIPTION:
There is considerable interest in E-Cs at the moment and the study would provide information on whether the E-C surpasses the tried and tested nicotine inhalator. If so, it would open a possibility of its utilization in smoking cessation, and provide encouragement for further examination of the role of sensorimotor replacements in the treatment of tobacco dependence.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers smoking at least 12 cigarettes per day
* First cigarette smoked within 60 minutes of waking up
* Willing to abstain from smoking for one day in 2 consecutive weeks.

Exclusion Criteria:

* Under 18 years of age
* Current psychiatric illness
* Pregnant or breastfeeding
* Enrollment in other research projects
* Used electronic cigarette and/or nicotine inhalator before

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hayden J McRobbie, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Tobacco Dependence Research Unit, London, United Kingdom

REFERENCES:
- [Background] West R, Hajek P. Evaluation of the mood and physical symptoms scale (MPSS) to assess cigarette withdrawal. Psychopharmacology (Berl). 2004 Dec;177(1-2):195-9. doi: 10.1007/s00213-004-1923-6. Epub 2004 Jun 4. PMID 15179542
- [Background] West RJ, Hajek P, Belcher M. Severity of withdrawal symptoms as a predictor of outcome of an attempt to quit smoking. Psychol Med. 1989 Nov;19(4):981-5. doi: 10.1017/s0033291700005705. PMID 2594893
- [Background] Cappelleri JC, Bushmakin AG, Baker CL, Merikle E, Olufade AO, Gilbert DG. Multivariate framework of the Brief Questionnaire of Smoking Urges. Drug Alcohol Depend. 2007 Oct 8;90(2-3):234-42. doi: 10.1016/j.drugalcdep.2007.04.002. Epub 2007 May 7. PMID 17482773
- [Background] Rose JE, Behm FM, Westman EC, Bates JE, Salley A. Pharmacologic and sensorimotor components of satiation in cigarette smoking. Pharmacol Biochem Behav. 2003 Sep;76(2):243-50. doi: 10.1016/j.pbb.2003.07.002. PMID 14592675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Tobacco Dependence Research Unit in London between January 2013 and February 2013.
Pre-assignment Details: Inclusion Criteria Smoking at least 12 cigarettes per day; first cigarette smoked within 60 mins of waking; willing to abstain from smoking for one day in 2 consecutive weeks.
  Exclusion Criteria Under 18s; current psychiatric illness; planning pregnancy, pregnant or breastfeeding; enrolled in other research; used EC or inhaler before.
Groups:
- Electronic Cigarette Then, Nicotine Inhalator: Randomised to receive electronic cigarette at the first session. Tested at study session then given to use ad-lib over 24 hours. Participants then returned to the clinic.
  1 week wash out period.
  Asked to return to clinic to receive Nicotine Inhalator. Tested at clinic then given product to use ad-lib over 24 hours. Participants then returned to the clinic.
  Nicotine: Inhalation of nicotine.
- Nicotine Inhalator Then, Electronic Cigarette: Randomised to receive Nicotine Inhalator at the first session. Tested at study session then given to use ad-lib over 24 hours. Participants then returned to the clinic.
  1 week wash out period.
  Asked to return to clinic to receive electronic cigarette. Tested at clinic then given product to use ad-lib over 24 hours. Participants then returned to the clinic.
Period: Overall Study
Arm/Group | Electronic Cigarette Then, Nicotine Inhalator | Nicotine Inhalator Then, Electronic Cigarette
Started | 28 | 23
Completed | 28 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was randomised crossover trial
Groups:
- Electronic Cigarette First, Then Nicotine Inhalator: Randomised to receive electronic cigarette at the first session. Tested at study session then given to use ad-lib over 24 hours. Participants then returned to the clinic.
  1 week wash out period.
  Asked to return to clinic to receive Nicotine Inhalator. Tested at clinic then given product to use ad-lib over 24 hours. Participants then returned to the clinic.
- Nicotine Inhalator First, Then Electronic Cigarette: Randomised to receive Nicotine Inhalator at the first session. Tested at study session then given to use ad-lib over 24 hours. Participants then returned to the clinic.
  1 week wash out period.
  Asked to return to clinic to receive electronic cigarette. Tested at clinic then given product to use ad-lib over 24 hours. Participants then returned to the clinic.
- Total: Total of all reporting groups
Arm/Group | Electronic Cigarette First, Then Nicotine Inhalator | Nicotine Inhalator First, Then Electronic Cigarette | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 22 | 48
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Comparison of E-C and Inhalator in Effects on Withdrawal Over 24 Hours of Use.
Description: Mood and Physical Symptoms Scale (MPSS): Measure of severity of urges to smoke and tobacco withdrawal symptoms.
  A five-point scale is used to rate 'How much of the time have you felt the urge to smoke in the past week?' ((1) 'not at all' to (5) 'almost all of the time') and 'How strong have the urges been?' ('no urges' to 'very strong'). Clients also rate depression, irritability, restlessness, hunger, poor concentration, poor sleep at night, and anxiety during the past week ((1)=not at all to (5)=extremely). The combined score to questions on depression, irritability, restlessness, hunger, and poor concentration are averaged to give the MPSS score. A higher score means a more severe rating of withdrawal.
  The primary outcome is a change in MPSS score between baseline and 24 hours (value at 24 hours minus value at baseline). Therefore, a smaller change in MPSS score represents a smaller increase in tobacco withdrawal symptoms.
Time Frame: 24 hours
Population: Reporting group
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Electronic Cigarette; Nicotine Inhalator: All study participants.
Arm/Group | Electronic Cigarette | Nicotine Inhalator
Number analyzed (Participants) | 51 | 51
units on a scale | 0.73 (0.64) | 0.86 (0.73)
Statistical Analysis 1: Comparison: Electronic Cigarette vs Nicotine Inhalator; Test type: Superiority; p = 0.17, t-test, 2 sided

2. Secondary Outcome: Change in Salivary Cotinine Levels After 24-hour Use.
Description: Cotinine is a measure sensitive enough to detect effects of a switch to different nicotine products and salivary cotinine was shown to be dependent on nicotine mouth exposure.
  The results show the mean change in salivary cotinine in each study arm (all study participants).
Time Frame: 24 hours
Population: Reporting group
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Electronic Cigarette | Nicotine Inhalator
Number analyzed (Participants) | 49 | 49
ng/ml | -66.32 (94.84) | -53.8 (119.4)
Statistical Analysis 1: Comparison: Electronic Cigarette vs Nicotine Inhalator; Test type: Superiority; p = 0.43, t-test, 2 sided

3. Secondary Outcome: Reinforcing Effects of Smoking
Description: Modified Cigarette Evaluation Questionnaire (mCEQ): Measure of reinforcing effects of smoking (pleasant feeling). Mean pleasant feeling from using product (rating 0-4). Higher value indicating the higher rating of pleasure.
Time Frame: 24 hours
Population: Reporting group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Electronic Cigarette | Nicotine Inhalator
Number analyzed (Participants) | 51 | 51
units on a scale | 2 (1.11) | 0.67 (0.89)
Statistical Analysis 1: Comparison: Electronic Cigarette vs Nicotine Inhalator; Test type: Superiority; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Airway Sensations
Description: Sensory effects: Measure of airway sensations (throat and chest). Mean enjoyment score (rating 0-4), higher the score indicating increased enjoyment.
Time Frame: 24 hours
Population: Reporting group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Electronic Cigarette | Nicotine Inhalator
Number analyzed (Participants) | 51 | 51
units on a scale | 1.65 (1.05) | 0.51 (0.7)
Statistical Analysis 1: Comparison: Electronic Cigarette vs Nicotine Inhalator; Test type: Superiority; p = 0.001, t-test, 2 sided

5. Secondary Outcome: Product Satisfaction
Description: Product satisfaction: Ratings of product satisfaction (when compared to cigarettes). Rating 0-4, with higher value indicating higher satisfaction ratings.
Time Frame: 24 hours
Population: Reporting group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Electronic Cigarette | Nicotine Inhalator
Number analyzed (Participants) | 51 | 51
units on a scale | 1.18 (1.05) | 0.59 (1.1)
Statistical Analysis 1: Comparison: Electronic Cigarette vs Nicotine Inhalator; Test type: Superiority; p = 0.003, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 hours after product use
Description: Adverse effects questionnaire (adapted from Hajek et al, 1989)
Groups:
- Electronic Cigarette; Nicotine Inhalator: All study participants used product.
Arm/Group | Electronic Cigarette | Nicotine Inhalator
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 30/51 | 34/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electronic Cigarette (N=51) | Nicotine Inhalator (N=51)
Dyspnoea (Cardiac disorders) | 8 (8) | 6 (6)
Dyspnoea at rest (Cardiac disorders) | 5 (5) | 2 (2)
Chest pain (Cardiac disorders) | 6 (6) | 4 (4)
Chest discomfort (Cardiac disorders) | 7 (7) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 18 (18)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 9 (9)
Dizziness (Nervous system disorders) | 9 (9) | 9 (9)
Headache (Nervous system disorders) | 10 (10) | 9 (9)
Sleep disturbance (Nervous system disorders) | 7 (7) | 5 (5)
Visual impairement (Eye disorders) | 4 (4) | 2 (2)
Disturbances in attention (Psychiatric disorders) | 9 (9) | 15 (15)
Nausea (Gastrointestinal disorders) | 7 (7) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes